CLINICAL TRIAL: NCT01079533
Title: Initiation of Colon Cancer Screening in Veterans
Brief Title: Initiation of Colon Cancer Screening in Veterans or "Start Screening Now"
Acronym: SSN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Duke University (Other); Boston University (Other)
Responsible Party: Principal Investigator, Sally Vernon, Professor - Health Promotion and Behavioral Science, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: R01CA112223-01A2 (NIH)
Record Dates: First submitted 2010-02-26; First posted 2010-03-03 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Neoplasms; Mass Screening; Patient Compliance; Intervention Studies; Clinical Trial
MeSH Terms: conditions — Colorectal Neoplasms; Patient Compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): A survey-only control arm will be compared to the experimental arm to determine whether the 3 different delivery channels are equally efficacious and cost-effective.
  Interventions: Behavioral: Control
- Minimal Cue and TLC (Experimental): Participants randomized to the experimental arm will receive a minimal cue after completing the baseline survey. A follow up survey will be sent 9 months after completion of the minimal cue to assess whether the participant received CRCS. If the participant has not had CRCS they will receive a more intensive telephone linked communication intervention. A second follow up will be sent 9 months after the TLC is delivered to assess final screening status.
  Interventions: Behavioral: Stepped CRCS Interventions

INTERVENTIONS:
Behavioral: Stepped CRCS Interventions — In Step 1, we will evaluate a theory-based minimal cue delivered by a letter, telephone call, or automated telephone call. Persons who do not complete CRCS in Step 1 will be randomized to Step 2 using principles of Motivation Interviewing. Step 2 also will determine whether an automated approach, telephone-linked communication (TLC), is as effective as a telephone counselor in promoting initiation of CRCS. Steps 1 and 2 together will address the important issue of the "dose" needed to encourage completion of CRCS.
  Other Names: Start Screening Now
  Arms: Minimal Cue and TLC
Behavioral: Control — A survey-only control arm will be compared to the experimental arm to determine whether the 3 different delivery channels are equally efficacious and cost-effective.
  Arms: Control

SUMMARY:
Initiation of colon cancer screening in veterans is a theory-based stepped intervention to increase first time colorectal cancer screening (CRCS) among male and female veterans age 50 and over.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the 2nd leading cause of cancer deaths in the US and risk increases with age. Colorectal cancer screening (CRCS) offers the possibility of both early detection and prevention. For those at average risk, CRCS beginning at age 50 is recommended. However, awareness and use of CRCS tests are low. We propose to conduct a randomized controlled trial to develop and test stepped interventions to increase initial uptake of CRCS in a nationally-representative, ethnically-diverse sample of male and female veterans. Our specific aims are to: (1) develop and pre-test stepped intervention components that are theory and evidence-informed; (2) implement and evaluate the process, efficacy, and cost-effectiveness of stepped interventions to increase an initial CRCS among male and female veterans aged 50-64 years; and (3) analyze the association between predictor variables and CRCS initiation and the mediating and moderating effects of the interventions, after each step. In Step 1, we will evaluate a theory-based minimal cue delivered by a letter, telephone call, or automated telephone call compared with a survey-only control group to determine whether the 3 different delivery channels are equally efficacious and cost-effective. Minimal cues are a cost-effective method that prompts to action those more willing to change and are easy to disseminate in real-world settings. Persons who do not complete CRCS in Step 1 will be randomized in Step 2 to more intensive interventions that address resistance. In Step 2 we will determine whether a theory-based, tailored telephone intervention, using principles of Motivation Interviewing, is effective when delivered as part of a sequential intervention process in which early adopters have been removed from the population. Step 2 also will determine whether an automated approach, telephone-linked communication (TLC), is as effective as a telephone counselor in promoting initiation of CRCS. Steps 1 and 2 together will address the important issue of the "dose" needed to encourage completion of CRCS. After each step, we will examine the mediating and moderating effects of the intervention to identify determinants of completion. For cancer screening intervention research to have the broadest public health impact, interventions must have the potential for dissemination. We designed our trial to move us toward the goal of disseminable interventions with evidence of external validity.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female Veteran age 50 to 64

Exclusion Criteria:

* Prior CRCS
* History of colon or bowel cancer, Crohn's disease, ulcerative colitis
* History of colon polyps
* Currently active duty military
* Outside of age range

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1892 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2011-11-03 (Actual); Study Completion 2014-07-31 (Actual)

PRIMARY OUTCOMES:
Colorectal Cancer Screening | 9 month follow up
  The primary outcome for the intervention trial is completion of an initial CRCS with 1 of the 5 currently recommended tests or test combinations. There will be one follow up measurement after each intervention step to assess whether uptake of CRCS was completed. The first measure is 9 months after the 1st intervention step. The second is 9 months after the 2nd intervention step.

CONTACTS AND LOCATIONS:
Overall Officials: Sally W Vernon, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston School of Public Health, Houston, Texas, United States